CLINICAL TRIAL: NCT05002647
Title: Relationship Between the Clinical Pharmacist & Antibiotic Use in Selected Infectious Disease Hospitals in El Beheira by Using the Electronic Program, Retrospective Cohort
Brief Title: Relationship Between the Clinical Pharmacist & Antibiotic Use by Using the Electronic Program
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Collaborators: Ministry of Health and Population, Egypt (Other Government)
Responsible Party: Sponsor
Other Study IDs: 14-2021/13
Record Dates: First submitted 2021-08-07; First posted 2021-08-12 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2021-08

CONDITIONS: Clinical Pharmacists; Electronic Medical Record
Keywords: clinical pharmacist; antibiotic consumption; antibiotic use; cost-saving

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- exposure group: Data from electronic clinical pharmacist records of two infectious disease hospitals
  Interventions: Other: NO intervention
- Non-exposure group A: Data from medical records of the hospital with no clinical pharmacy.
  Interventions: Other: NO intervention
- Non-exposure group B: Data from a medical record of the hospital with clinical pharmacy, but the department did not cover by the clinical pharmacy
  Interventions: Other: NO intervention

INTERVENTIONS:
Other: NO intervention — There is no intervention

SUMMARY:
A retrospective cohort study to explore the association between clinical pharmacists' interventions and antibiotic consumption through the use of the medical electronic reports and to identify mortality and cost savings in hospital infectious disease.

DETAILED DESCRIPTION:
The role of clinical pharmacist includes :

1. a check of suitable selection and dosing of antimicrobials according to the diagnosis, type of infection, antimicrobial cultures as possible, comorbidities of patients (renal or hepatic function, etc), adverse effect, and drug interaction with other drugs.
2. Documentation of the clinical intervention, cost-saving, adverse effect,, antimicrobial culture and antimicrobial consumption on the electronic program (CPC "clinical patient care").
3. The clinical pharmacist inspector reviews the data recorded on CPC.

ELIGIBILITY:
Inclusion Criteria:

* All inpatient with infectious disease (disorders caused by organisms as (bacteria, viruses, fungi, or parasites).

Exclusion Criteria:

* Any other cause of hospital admission other than infectious disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who administered antimicrobials
Sampling Method: Probability Sample
Enrollment: 2601 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Antimicrobial consumption | 2 years
  consumption of antimicrobials (defined daily doses / 100 patient-days)
Days of therapy (DOT) | 2 years
  Number of days of each antimicrobial received for therapy
Length of therapy(LOT) | 2 years
  The number of days a patient takes an antibacterial drug, regardless of the number of different medications

SECONDARY OUTCOMES:
cost savings | 2 years
  (initial treatment cost × days before intervention) - (cost after intervention × days with this treatment),
Mortality rate | 2 years
  in-hospital mortality rate (%)
Antimicrobial resistance | 2 years
  resistance defined as resistance to at least one antimicrobial from the panel for all organisms, and for a subset of organisms belonging to the ESKAPE group (Enterococcus faecium, S. aureus, Klebsiella pneumonia, Acinetobacter baumannii, Pseudomonas aeruginosa , and Enterobacter spp.
The incidence of adverse reaction of antimicrobial | 2 years
  An unexpected medical problem that happens during treatment with antimicrobial.

CONTACTS AND LOCATIONS:
Overall Officials: Amira zidane, Principal Investigator — Ministry of Health and Population, Egypt
Locations (1):
- Ministers of health, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Karakonstantis S, Kalemaki D. Antimicrobial overuse and misuse in the community in Greece and link to antimicrobial resistance using methicillin-resistant S. aureus as an example. J Infect Public Health. 2019 Jul-Aug;12(4):460-464. doi: 10.1016/j.jiph.2019.03.017. Epub 2019 Apr 10. PMID 30981652
- [Background] Dyar OJ, Huttner B, Schouten J, Pulcini C; ESGAP (ESCMID Study Group for Antimicrobial stewardshiP). What is antimicrobial stewardship? Clin Microbiol Infect. 2017 Nov;23(11):793-798. doi: 10.1016/j.cmi.2017.08.026. Epub 2017 Sep 4. PMID 28882725
- [Background] Ourghanlian C, Lapidus N, Antignac M, Fernandez C, Dumartin C, Hindlet P. Pharmacists' role in antimicrobial stewardship and relationship with antibiotic consumption in hospitals: An observational multicentre study. J Glob Antimicrob Resist. 2020 Mar;20:131-134. doi: 10.1016/j.jgar.2019.07.009. Epub 2019 Jul 16. PMID 31323427